## Official Title of the Study:

Comparative Clinical Evaluation of Partial Coverage CAD/CAM Restoration Versus Nanohybrid Composite of Carious Hypomineralized Permanent Molars: A Randomized Controlled Trial

NCT Number: Not yet assigned

**Date of the Document:** December 2023

# Comparative Clinical Evaluation of Partial Coverage CAD/CAM Restoration Versus Nanohybrid Composite of Carious Hypomineralized Permanent Molars: A Randomized Controlled Trial.

التقييم السريري المقارن للتغطية الجزئية لترميم CAD/CAM مقابل مركب Nanohybrid من الأضراس الدائمة ناقصة المعادن: تجربة عشوائية محكومة.

| | | Protocol checklist | D 1 | D |
|---|---|---|---|---|
| Section and topic | Item no. | Checked item | Reported on page No. | Reviewer's check |
| | 1 | Title | | |
| I. Administrative information | 2 | Protocol registration | | |
| | 3 | Protocol version | | |
| | 4 | Funding | | |
| | 5 | Roles and responsibilities | | |
| II. Introduction | | | | |
| | 6 a | Research question | | |
| | | Statement of the problem | | |
| A) Background and Rationale | | Rationale for carrying out the trial | | |
| | | Review of literature | | |
| | 6 b | Choice of comparators | | |
| | | Aim of the study | | |
| B) Objectives | 7 | Hypothesis | | |
| | | Primary and secondary objectives | | |
| C) Trial design | 8 | Trial design | | |

| III. Methods | | |
|---|---|---|
| | 9 | Study setting |
| | 10 | Eligibility criteria |
| A) Participants, interventions | 11 | Interventions |
| & outcomes | 12 | Outcomes |
| a dutcomes | 13 | Participant timeline |
| | 14 | Sample size |
| | 15 | Recruitment |
| B) Data collection, management, | 16 | Data collection methods |
| and analysis | 17 | Data management |
| | 18 | Statistical methods |
| | 19 | Data monitoring |
| C) Monitoring | 20 | Harms |
| | 21 | Auditing |
| | 22 | Research ethics approval |
| | 23 | Protocol amendments |
| | 24 | Informed Consent |
| IV. Ethics and dissemination | 25 | Confidentiality |
| | 26 | Declaration of interests |
| | 27 | Access to data |
| | 28 | Ancillary and post-trial care |
| | 29 | Dissemination policy |

| | Re | search plan committee | |
|----------------|-----------------|-----------------------------|------|
| 2. | | | |
| 1. | | | |
| Name | | Signature | Date |
| | <b>Evidence</b> | based committee (Reviewers) | |
| VI. References | | | |
| | 31 | Biological specimens | |
| V. Appendices | 30 | Informed consent materials | |

| Name | Signature | Date |
|------|-----------|------|
| 1. | | |
| 2. | | |

#### **Administrative information:**

#### 1. Title:

Comparative Clinical Evaluation of Partial Coverage CAD/CAM Restoration Versus Nanohybrid Composite of Carious Hypomineralized Permanent Molars: A Randomized Controlled Trial.

- 2. Protocol Registration:
- 3. Protocol version:
- 4. Funding: Self-funded

University Responsibilities: All contribute in initiated the study design, will generate random sequence, contribute in clinical work, provide statistical expertise in clinical trial design and make the final edited of the article.

#### II. Introduction:

#### 5. Background and rationale:

Hypomineralization of carious permanent molars is defined as qualitative defects caused by disruptions in either the calcification or maturation phases of amelogenesis. (1)

#### **Statement of the problem:**

Conventionally, stainless steel crowns were used for those molars. However, due to the need for esthetics and the young age of patients, it was necessary to look for a cosmetic and conservative restoration alternative. (2) Partial coverage restorations were recommended as a substitute for crowns to maintain teeth healthy. It is considered a minimally invasive approach. (3)

#### The rationale for conducting the research:

Conventional restoration for such hypomineralized molars necessitates massive removal of the tooth structure to receive full coverage crowns that cause more biologically harmful consequences like pulp exposure especially in young permanent teeth and aggressive tooth structure loss (4). To fulfill the biological criteria for tooth preparation, conservatism is the major notion and goal that dental practitioners strive to achieve. Nowadays, minimally invasive techniques are frequently employed to

support this idea. To meet the growing need for conservative and esthetics tooth restorations, partial

coverage ceramic restorations are becoming more necessary. These CAD/CAM restorations show

satisfactory mechanics, restoring function, and esthetic with preserving tooth structure (5)

Since all materials used to treat such cases have distinct chemical compositions, they have

different properties that affect their clinical outcome. Therefore, it is essential to compare them clinically

because any restoration's clinical outcome affects its long-term success. According to the null

hypothesis, different materials would not significantly affect the clinical result of ceramic overlay

restorations.

Patients in all groups will receive a minimally invasive restoration with high esthetic advantages

(Protection of the weak cusps and elimination of carious lesions with an esthetic way out) and long-term

success of their affected carious hypomineralized permanent molars (IPS e.max CAD or Direct

nanohybrid flowable composite) that require minimal preparation depends on the type of restoration will

receive.

Aim of the study:

This randomized controlled trial study will evaluate the clinical success of direct nanohybrid flowable

composite versus IPS e.max CAD Partial Coverage.

**Research question:** 

Are the direct nanohybrid flowable composite and IPS e.max CAD Partial Coverage clinically successful

materials in restoring the carious Hypomineralized Permanent Molars?

**PICOS:** 

**P:** Patients suffer from hhypomineralized permanent molars

I: Direct nanohybrid flowable composite

C: IPS e.max CAD

O: Clinical Success (aesthetics, functional and biological criteria))

**II. Methods** 

**Study Design:** 

Study design: Randomized Controlled Trial

Estimated Enrolment: 48 Carious Hypomineralized Permanent Molars

Allocation: Randomized

Intervention Model: Parallel Assignment

Primary Purpose: Restorations Hypomineralized Permanent Molars

5

Official Title: Comparative Clinical Evaluation of Partial Coverage CAD/CAM Restoration Versus Nanohybrid Composite of Carious Hypomineralized Permanent Molars: A Randomized Controlled Trial.

Estimated Study Start Date: December 2023 [Time frame: 12 months] Estimated Primary

Completion Date: January 2025

#### Trial design:

The study is a randomized controlled trial (RCT) where 2 arm parallel groups with a 1:1 allocation ratio were compared. The child participants and the legal guardian of each participating child and the statistician were blinded.

#### **Outcome Measures:**

- 1. **Primary outcome:** Clinical success [Time Frame: 12 months].
  - According to FDI World Dental Federation criteria [Appendix A]
  - There were three assessment categories (aesthetics, function, and biological), each with five subcategories. From best to worst, the subcategories were:
    - (1) clinically excellent, (2) clinically good, (3) clinically sufficient, (4) clinically not sufficient but repairable, and (5) clinically unacceptable. Assessment with category (5) was rated as a clinical failure.
  - At the follow-up visits over one year at (baseline "1 day ", 6 and 12 months) after cementation., will take standardized photographs and the restorations will clinically evaluate by an independent and calibrated clinician.

#### **Eligibility Criteria**

Ages Eligible for Study: Above 6 Years

Sexes Eligible for Study: All

Accepts Healthy Volunteers: Yes

#### Criteria

#### **Inclusion Criteria:**

- 1. Above 6 years old
- 2. Cooperative children with large carious First Permanent Molars (FPM) lesions associated with weak cusps and defected hypo-mineralized enamel.
- 3. Apparently healthy patients.
- 4. Patients will be available to be clinically reviewed up to 1 year

#### **Exclusion Criteria:**

- 1. Patients with Symptoms of pulpitis.
- 2. Patients with uncontrolled active tooth decay or periodontal disease (i.e. 4+ mm probing depth and bleeding on probing).
- 3. Poor oral hygiene and motivation.
- 4. Patients with parafunctional habits (e.g., bruxism, biting on hard objects).
- 5. Patients with debilitating illnesses or complicating medical conditions

#### **Explanation regarding the choice of comparators:**

**IPS e.max CAD**: Till now, glass—ceramic-based restorations still offer the best translucency and esthetic qualities. The novel generation of lithium disilicate-based materials as IPS e.max CAD provides standard thickness and quick fabrication. Moreover, the adhesive technique used with this restoration type significantly raises its mechanical properties. (6)

**Beautifil Flow Plus X** (Shofu)is a bioactive flowable nano-hybrid restorative with a newly developed patented nanofiller. It is indicated for all classes including occlusal and cusp. It has all the Giomer Technology attributes, anti-bacterial, acid neutralization, and fluoride release and recharge, with improved handling and effortless polishing, and maintains a long-lasting shine. Beautifil Flow Plus X has the strength, durability, and aesthetics of a hybrid composite. (7)

#### Sample size (Power analysis):

Sample size calculated depending on a previous study (Alaa M. Eldehna a et al., 2023) as reference. (8) According to this study, the probability of surface gloss as an aesthetics criterion in group 1 is 0.96. If the estimated probability of group 2 is 0.6, we will need to study 20 cases in each group with probability (power) 0.8. The Type I error probability. We used the chi-squared test to evaluate that was performed by using P.S.Power 3.1.6. Total sample size increased to 24 subjects per group to compensate for a 15 % drop out. Sample size calculation was achieved using chi-squared test to evaluate that was performed by using P.S. Power3.1.6, software Version 3.1.2 (Vanderbilt University, Nashville, Tennessee, USA).

#### **Statistical Methods**

#### **Statistical analysis:**

Data was collected, tabulated, and statistically analyzed using Microsoft Excel ® 2016, Statistical Package for Social Science (SPSS)® Ver. 24. And Minitab ® statistical software Ver. 16.

#### Handling of numerical / quantitative variables:

Numerical data will be explored for normality by checking the data distribution using Kolmogorov-Smirnov and Shapiro-Wilk tests. Data will be presented as mean & amp, standard deviation. If data will be normally distributed comparison between 2 different groups will be performed by using independent t-test, comparison between 2 related groups will be performed by using Paired t-test, while comparison between more than 2 groups will be performed by using One Way ANOVA test followed by Tukey's Post Hoc test for multiple comparisons. If data will be non-parametric data comparison between 2 different groups will be performed by using Mann-Whitney test, comparison between 2 related groups will be performed by using Wilcoxon Signed Rank test, while comparison between more than 2 groups will be performed by using Kruskal-Walli's test.

#### Handling of categorial / qualitative variables:

Data will be presented as frequency and percentages. All comparisons will be performed by using Chi square test.

#### **Recruitment:**

The study will be conducted at the pediatric dentistry department of MSA University pediatric outpatients. All subjects will be monitored and reviewed at day 1 after 6 months and 12 months.

#### Post-trial care

- · Oral hygiene instructions and serving brush and toothpaste
- Dietary recommendations

#### **Patients Guardians Consent and Ethical Approval**

An informed Consent will be read in detail, explained and signed by the patients' guardians and will make sure that all risk expectations are well understood along with benefits and expected outcomes of this clinical research trial to the patient's well-being. The consent will authorize a treatment plan aimed at a mutually acknowledged treatment goal.

#### [Appendix B]

#### **Ethical Approval Number:**

#### **III. References**

- Dhareula A, Goyal A, Gauba K, Bhatia SK, Kapur A, Bhandari S. A clinical and radiographic investigation comparing the efficacy of cast metal and indirect resin onlays in rehabilitation of permanent first molars affected with severe molar incisor hypomineralisation (MIH): a 36-month randomised controlled clinical trial. European Archives of Paediatric Dentistry. 2019 Oct;20:489-500.
- 2. De Leon, F.M., Garza, N., Coronado, J., Ancona, M., 2022. Indirect ceramic overlay restorations as a minimally invasive alternative for posterior rehabilitation. Inter. J. App. Dent. Sci. 8, 79–83.
- 3. Schiffenhaus, S., 2021. The Nonretentive Ceramic Overlay. A biomimetic alternative to the full coverage crown. Ins. Dent. J. 17, 24–31.
- 4. Linner, T., Khazaei, Y., Bu"cher, K., Pfisterer, J., Ku"hnisch, J., 2020. Comparison of four different treatment strategies in teeth with molar-incisor hypomineralization-related enamel breakdown—A retrospective cohort study. Int. J. Paediatr. Dent. 30, 597–606.
- Mohammed, Z., Majeed, M., 2020. Effect of cementation protocol on the marginal adaptation of indirect overlay restorations fabricated from two different all-ceramic CAD/CAM materials. J. Res. Med. Dent. Sci. 8, 518–525.
- 6. Phark JH, Duarte Jr S. Microstructural considerations for novel lithium disilicate glass ceramics: A review. Journal of Esthetic and Restorative Dentistry. 2022 Jan;34(1):92-103.
- 7. Pinto NS, Jorge GR, Vasconcelos J, Probst LF, De-Carli AD, Freire A. Clinical efficacy of bioactive restorative materials in controlling secondary caries: a systematic review and network meta-analysis. BMC Oral Health. 2023 Dec;23(1):1-20.

8. Eldehna AM, Montaser AG, ALrafee SA, Abdelgawad A. Clinical outcome of CAD/CAM overlays of MIH affected young permanent molars. The Saudi Dental Journal. 2023 Sep 1;35(6):699-706.

## Appendices

Appendix A: FDI World Dental Federation criteria

| Properties | Parameters | Excellent<br>Score1 | Good<br>Score 2 | Satisfactory<br>Score 3 | Mediocre<br>Score 4 | Poor<br>Score 5 |
|---|---|---|---|---|---|---|
| Esthetic | Surface<br>lustre | Luster comparable to enamel | Slightly dull;<br>some isolated<br>pores | Dull surface;<br>multiple pores<br>(>1/3 of the<br>surface) | Rough surface;<br>presence of voids | Very rough surface |
| | Marginal<br>and Surface<br>staining | No staining | Minor staining | Moderate staining | Pronounced staining | Severe<br>staining |
| | Anatomical form | Ideal form | Form slightly deviated | Moderate changes of form | Pronounced changes of form | Lost of form |
| Functional | Fracture of<br>material and<br>retention | No fractures or cracks | Small hairline<br>cracks | Two or more<br>larger hairline<br>cracks and/or<br>chipping (not<br>affect marginal<br>integrity) | Chipping<br>fractures, bulk<br>fractures with<br>or without<br>partial loss (less<br>than half of the<br>restoration) | Partial or<br>compete<br>loss of<br>restoration |
| | Marginal<br>adaptation | Harmonious<br>outline,<br>no gaps | Marginal gaps<br>(<150 μm);<br>small marginal<br>fractures | Marginal gaps<br>(>150 μm and<br><250 μm);<br>several marginal<br>fractures | Marginal<br>gaps >250<br>μm or dentin/<br>base exposed;<br>severe marginal<br>fractures | Restoration<br>lost but<br>in situ;<br>generalized<br>major gaps |
| | Radiographic examination* | No pathology | Adhesive pooling and/or slightly internal maladjustment of the restoration | | Evidence of secondary caries;<br>apical pathology; fracture or loss<br>of restoration or tooth | |
| Biological | Postoperative<br>(hyper)<br>sensitivity<br>and tooth<br>vitality | No<br>hypersensitivity;<br>normal vitality | Minor<br>hypersensitivity<br>for a limited<br>period of time<br>(<1 week);<br>normal vitality | Moderate hypersensitivity for a limited period of time (>1 week and <6 months); mild sensitivity, no complains | Intense<br>hypersensitivity;<br>cold sensitivity<br>with minor<br>subjective<br>symptoms | Acute pulpitis<br>or non<br>vital tooth;<br>endodontic<br>treatment is<br>mandatory |
| | Recurrence of caries | No secondary or primary caries | Small and<br>localized<br>demineralization<br>area | Larger areas of<br>demineralization<br>with no dentin<br>exposure | Localized and accessible caries with cavitation | Deep<br>secondary<br>caries with<br>exposed dentin |
| | Tooth<br>integrity | Complete integrity | Small marginal<br>enamel fracture<br>(<150 µm);<br>hairline crack in<br>enamel | Marginal enamel<br>fractures (<250<br>μm); multiple<br>cracks | Major marginal<br>enamel fractures<br>(>250 μm) with<br>exposed dentin;<br>large enamel<br>chipping or wall<br>fracture | Cusp or tooth fracture |
| | Adjacent<br>mucosa | Healthy mucosa<br>adjacent to<br>restoration | Healthy mucosa<br>after minor<br>removal of<br>mechanical<br>irritation | Alteration of<br>mucosa but<br>not suspicion<br>of causal<br>relationship<br>with restorative<br>material | Suspected mild<br>allergic lichenoid<br>or toxic reaction | Suspected<br>severe allergic<br>lichenoid or<br>toxic reaction |

# [Appendix B]: Informed consent

#### \_Scientific Research Ethics Committee

Informed Consent for Volunteers

#### **Research Title:**

Comparative Clinical Evaluation of Partial Coverage CAD/CAM Restoration Versus Nanohybrid Composite of Carious Hypomineralized Permanent Molars: A Randomized Controlled Trial

#### Objective of the Research:

This randomized controlled trial study will evaluate the clinical success of direct nanohybrid flowable composite versus IPS e.max CAD Partial Coverage.

# **Introduction and Details of What Will Be Performed on the Patient** (Work plan)

- Direct benefit to the volunteer

[] Verbal explanation

- Scientific benefits and general expected benefits from the research
- Side effects, risk level, expected occurrences, and how to handle them
- Patient duties regarding oral and dental health care during the research/study

| [] Full understanding of the patient regarding the research steps: |
|--------------------------------------------------------------------|
| [] Reading |

I have carefully reviewed and understood the purpose of the research and the nature of this study. I understand what is required to complete these procedures.

- 1. The research doctor has informed me of possible alternative treatments to this research.
- 2. The research doctor has informed me of all potential risks of this research and how to handle them.
- 3. I agree to photography, recording, and all types of radiographs required in this study, provided that my identity will not be disclosed.
- 4. I have provided an accurate report about my health history. I have informed the doctor of all types of health reactions or unusual allergies to medications, foods, insect stings, anesthetics, dust, or any other materials, or abnormal bleeding, or any other conditions related to my health.
- 5. I declare that I am not participating in any other research from the start of this study until its end, and I will inform the research doctor if I participate in any other research during this study.
- 6. I pledge to return any medical equipment (tools) used in the research if I stop or upon completion of the research.

After being informed of the available information regarding the research, the volunteer or their guardian is free to choose whether or not to participate. If they agree, they are requested to fill in the data below, knowing that they have the right to withdraw from the research at any time without giving reasons, with due regard for the researcher's right to retrieve any medical devices or tools used for research purposes that are in the volunteer's possession (as required by the researcher).

| Volunteer's Name: |
|---|
| Date of Birth: |
| National ID (if available): |
| Guardians or companion's name (if applicable): |
| National ID: |
| Address: |
| Phone: |
| Date: |
| The physician responsible undertakes to maintain the confidentiality of the volunteer's information in |

The physician responsible undertakes to maintain the confidentiality of the volunteer's information in the research, mentioning the methods used for this, such as replacing names with coded numbers or hiding facial features in photographs where possible, etc.

#### Researcher's signature: